CLINICAL TRIAL: NCT06123689
Title: A Prospective, Randomized, Clinical Trial to Evaluate the Safety and Efficacy of AMT-RegeneraActiva in the Management of Knee Osteoarthritis (OA)
Brief Title: Safety and Efficacy of AMT-RegeneraActiva in the Management of Knee Osteoarthritis (OA)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Human Brain Wave S.r.l. (Industry)
Collaborators: Nextrasearch S.r.l.s. (Other); Ibismed S.r.l. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RE78.22.01
Record Dates: First submitted 2023-10-27; First posted 2023-11-09 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthritis
Keywords: knee osteoartrithis; knee chondropathy
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AMT-Regenera activa (Experimental): All the patients of the group will be treated with one unique articular injection of autologous micrografts obtained through the Rigenera® Technology
  Interventions: Device: AMT-Regenera activa
- Hyalubrix (Active Comparator): All the patients of the group will be treated with one unique articular injection of Sodium Hyaluronate (Hyalubrix 60 -1,5%-2ml vial)
  Interventions: Device: Hyalubrix

INTERVENTIONS:
Device: AMT-Regenera activa — Patient's preparation: is an ambulatory procedure, the sterility of the Micrograft and the method should be guaranteed during the whole procedure.
  Punch biopsy extraction:
  The punch should be obtained by the posterior auricular shell area. The zone cleaned with antiseptic solution. Anesthesia is applied in the posterior zone in the base area of the auricular shell. It should be applied superficially to separate the skin from the cartilage . Should be obtained by 3 dermic punches of 2,5mm diameter. The skin is separated from the perichondrium and cartilage.
  1. Once the samples are obtained, they must be put on the metallic grid of the Rigeneracon
  2. Afterwards, 4 ml of Saline solution are added in the inferior part of the Rigeneracon, then close the lid and then put it in the machine with the needed adaptors.
  3. The samples are processed for 6 minutes
  4. The Rigeneracon is extracted from the machine.
  Arms: AMT-Regenera activa
Device: Hyalubrix — Patients randomized in Group 2 Sodim Hyaluronate (Hyalubrix 60 -1,5%-2ml vial). NOTE: For the infiltration in the medial knee compartment treatment, the use of intramuscular needle is recommended.
  The care post-treatment The homeostasis of the donor's area is achieved by mechanical compression. Usually, there is no need of stitches.
  Often it can be seen a bit of inflammation during the first 24-72 hours. The use of analgesic drugs is recommended, avoiding the NSAID, they can interfere in the function of micrografts. Apply intermittently cold on the area or a compressive bandage, if needed
  Arms: Hyalubrix

SUMMARY:
The goal of this clinical trial is to compare in 60 patients suffering for Knee OA to demonstrate that AMT-RegeneraActiva is able to speed up the improvement process of knee osteoarthritis (OA) compared to Sodium Hyaluronate Participants will [describe the main tasks participants will be asked to do, treatments they'll be given and use bullets if it is more than 2 items].

Researchers will compare 2 Groups to see to demonstrate that AMT-RegeneraActiva is able to speed up the improvement process of knee osteoarthritis (OA) compared to Sodium Hyaluronate to pain management and improvement of functionality.

DETAILED DESCRIPTION:
All the patients participating in the study will have had been diagnosed with degenerative knee chondropathy from grade II to III of Kellgren-Lawrence grading scale and they will have signed a consent informed. The age rate established is from 25 to 65 years old. All the patients, except control group, will be treated with one unique articular injection of autologous micrografts obtained through the Rigenera® Technology. The control group will receive Sodium Hyaluronate (Hyalubrix 60 -1,5%-2ml vial). To assess the level of satisfaction of the patient, the reduction of pain, and the functional state of the articulation, Knee Osteoarthritis Outcome Score (KOOS) will be used, before the treatment, 3 months after the treatment, and at 6 months after the treatment.

The patients will be randomized as:

* Group (Arm) 1: AMT-RegeneraActiva
* Group (Arm) 2: Sodium Hyaluronate(Hyalubrix 60 -1,5%-2ml vial).

Patients in both treatment arms will be provided with paracetamol (500 mg/tablet) as rescue medication for relieving knee's pain. This will be taken as needed for pain with a maximum of 4 tablets or 2 grams of paracetamol per day up to 4 days per week.

If more rescue medication is needed for pain, (recorded as the 'Number of Rescue Medication Taken for pain' in the daily diary) the patient will be considered a treatment failure. Patients deemed treatment failures for rescue medication use will continue to participate in follow-up visits for safety.

During the study patients in both arms must report in a daily paper diary consumption of rescue medication, in particular, the following information will be collected:

Rescue paracetamol for OA:

* Amount of rescue medication taken for OA in the past 24 hours.
* Any non-rescue pain medication for OA or for pain other than OA

The consumption of rescue medication will be checked from the Investigators will be carefully documented at all visits during the study.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 25-65 inclusive with open physis confirmed by MRI (Size of the articular cartilage lesion is ≥ 2 cm2)
2. Documented symptomatic stable diagnosed degenerative knee chondropathy from grade II to III based on MRI without changes of osteoarthritis and no prior history of knee surgery. The MRI diagnosis must be within a 3-month time period prior to consent.
3. Joint pain: 20-mm - 60-mm on VAS (Visual Analog Scale) at the time of Screening
4. The patient must be able to hold still without sedation for approximately 1 hour and must pass MRI screening evaluation for retained metal.
5. Body Mass Index (BMI) ≤ 30 kg/m2 (extremely obese)
6. No meniscal surgery within the past 3 months and more than 5mm of meniscal rim remaining
7. Patient has complied with the requirements for rescue medication (no more than 4 tablets or 2 grams of paracetamol per day up to 4 days per week
8. Patients will have signed a consent informed

Exclusion Criteria:

1. Patients with polyarticular disease (not applicable to polyarticular disease of the knees as the most symptomatic knee will qualify for the study)
2. Patients with blood disorders (Blood disorders (thrombopathy, thrombocytopenia, anemia with hemoglobin <9g/dL).
3. Patients who had intra-articular treatment with steroids within 3 months
4. Patients who are pregnant or nursing at the time of consent.
5. Patients with inflammatory arthritic conditions (e.g. rheumatoid arthritis)
6. Patients who had previous knee surgery
7. Additional disabilities in any of the lower limbs that would interfere with any of the clinical assessments.
8. Chronic use of NSAID (defined as taking NSAID regularly every week for the last 6 months), steroids or chemotherapy drugs
9. Treatment with NSAIDs within 15 days prior to randomization in this study
10. Patients with a BMI over 30. Due to the fact that this study utilizes an injection technique which may be inaccurate in obese subjects.
11. Patients with acute or chronic renal failure
12. Patients who received a MRI diagnosis of OCD but do not have the specific cartilage imaging sequences.
13. Clinical or laboratory evidence of septicemia
14. Any problems in the ear tissue affecting the collection of cartilage

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
AMT Regenera improvement of pain management | 6 months overall
  To demonstrate that AMT-RegeneraActiva is able to speed up the change process of knee osteoarthritis (OA) compared to Sodium Hyaluronate (Hyalubrix 60 -1,5%-2ml vial) to pain management and consequent change of functionality in patients with knee OA (grade II-III Kellgren-Lawrence grading scale) from baseline after unique administration of ATM Regenera-Activa treatment by interarticular injection.
  KOOS score will be tool to measurement of this change

SECONDARY OUTCOMES:
IKDC improvement | 6 months overall
  IKDC patient reported SCORE

CONTACTS AND LOCATIONS:
Overall Officials: Vincenzo Salini, Prof. MD, Principal Investigator — Ospedale San Raffaele; Carlo Fiorentini, Prof. MD, Principal Investigator — Policlinico San Donato Milanese

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR
Time Frame: from within 6 months from the end, no limits of visibility